CLINICAL TRIAL: NCT06257524
Title: Improving Pediatric Readiness of Emergency Departments in Manitoba, Canada: a Randomized Controlled Trial and Survey Sampling
Brief Title: Pediatric Readiness Intervention in Manitoba
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other); Children's Hospital Research Institute of Manitoba (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Alex Aregbesola, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HS25688 (H2022:305)
Record Dates: First submitted 2023-10-11; First posted 2024-02-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Readiness
Keywords: Pediatric readiness, emergency department, Manitoba, RCT
MeSH Terms: conditions — Emergencies | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDIM component 1, 2, and 3 (Experimental): Intervention component 2 to be tested. Pediatric resources toolkits availability via Translating Emergency Knowledge for Kids network (TREKK). Investigators will provide resource toolkits to support clinical care in pediatric sepsis, seizure, diabetes ketoacidosis, dehydration, hypovolemic shock, and respiratory conditions.
  Intervention component 3 to be tested: Ongoing interactions, and intensive training and education sessions. Investigators will hold training and education sessions at the sites. These will include (a) One on-site training (for 4-4.5 hours) with simulation sessions.
  Interventions: Other: Education and training
- PDIM component 1 (Active Comparator): Customized report to the general EDs and discussion with the general EDs on the gaps identified. Investigators will discuss customized baseline WPRS with each general ED, including implications of the gaps identified relative to their local context and the general ED priorities (1.5hrs/session x 2).
  Interventions: Other: Education and training

INTERVENTIONS:
Other: Education and training — Pediatric resource toolkits availability via TREKK for Kids Ongoing interactions, and intensive training and education sessions

SUMMARY:
The goal of this clinical trial is to improve emergency care of children in Manitoba by increasing the weighted pediatric readiness scores (WPRS) of the general EDs through the implementation of provincially derived interventional measures (PDIM). Investigators want to test the effects of PDIM on the general EDs in Manitoba. The main questions it aims to answer are:

* What is the magnitude and direction of the effect of implementing PDIM on baseline WPRS of the general EDs, if any?
* Which implementation strategies effectively support the full incorporation of PDIM to increase the WPRS of general EDs across Manitoba? The participating general EDs will be asked to
* Gather individuals providing emergency care in their centers for training and education around PDIM.
* Select a lead person who will act as the general ED Champion.

DETAILED DESCRIPTION:
Description Investigators defined the inclusion and exclusion criteria using the PICO framework. They will implement a prospective single-blinded RCT involving 17 gEDs. The entire study will be coordinated at the Children's Hospital Research Institute of Manitoba. Investigators will assess for compliance in a scheduled pattern after the education and training sessions using a checklist. They will also sample all the 17 gEDs via RedCap link, post intervention.

PDIM is composed of 3 components. (1) Customized report to the gEDs and discussion with the gEDs on the gaps identified (1.5hrs/session x 2). (2) Pediatric resource toolkits availability via Translating Emergency Knowledge for Kids (TREKK). (3) Ongoing interactions, and intensive training (2.5hrs/session x 1) and education sessions. The gEDs in the control group will receive only the first component of the 3 components of PDIM.

Randomization Investigators have completed the randomization of anonymized 17 of the 28 gEDs. Randomization was performed using an R statistical software program into intervention (n=9) versus control (n=8), in a ratio of 1:1 within pairs. The gEDs were paired using a hierarchical cluster analysis based on the baseline WPRS, ED volume and ED location.

Survey The validated survey (n/100) will collect information around the six domains of the gEDs post intervention including coordination of patient care, ED staffing and training, quality improvement, patient safety, policies and procedures, and availability of pediatric equipment/supplies.

Data management and statistical analysis Phase 1 Frequentist approach - The investigators will perform a meta-analysis to generate a forest plot showing the mean change in WPRS of gEDs with 95% CI. The association between the change in WPRS and types of intervention will be examined in random-effects models.

Phase 2 & Phase 3 Frequentist approach - Investigators will perform a descriptive analysis on the baseline characteristics of participating gEDs. The difference in baseline characteristics of the gEDs between intervention and control groups will be assessed using Pearson χ2 or Fisher exact test for categorical data and t-test/Mann-Whitney U for continuous variables. The difference between the baseline WPRS and post intervention WPRS of the gEDs will be compared using paired-sample t-tests.

Bayesian approach - The intervention effect will be estimated using a vague prior called Cauchy, as will the other parameters in the fully Bayesian model. Investigators will report the posterior probability of a positive finding using a threshold effect size greater than 5, Pr(Effect > 0 | data), and also with an effect size greater than 7, Pr(Effect > 7 | data).

Sample size estimation - Investigators assumed an optimistic prior for the intervention effect to be a Cauchy distribution centered at 10, representing 80% certainty that the effect size is between 7 and 10.

Significance of research:

Implementing PDIM will help address the gaps identified in the gEDs in Manitoba. This study has the potential of increasing overall WPRS, which has been shown to have a strong inverse correlation with pediatric mortality. It will improve acute care for children regardless of the location of the gED in Manitoba.

ELIGIBILITY:
Inclusion Criteria: All criteria must be met.

* General ED located in Manitoba
* Offering emergency care to children aged 0-18 years during the study period
* Participated in the baseline evaluation of WPRS of the general EDs in Manitoba in 2019-2021

Exclusion Criteria:

* General EDs not providing emergency care to children aged 0-18 years during the study period.
* General EDs with no baseline WPRS

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Weighted Pediatric Readiness Scores | 9 months
  To be measured using the Manitoba Pediatric Readiness Initiative for Emergency department Survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada